CLINICAL TRIAL: NCT05949606
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety and Efficacy of SI-B001+SI-B003 With or Without Chemotherapy (SI-B001+SI-B003± Chemotherapy) in the Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of SI-B001+SI-B003± Chemotherapy in the Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001-SI-B003-202
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants will receive treatment during the first cycle. Participants with clinical benefits received more cycles of additional therapy. Administration will be discontinued due to disease progression or occurrence of intolerable toxicity or other reasons.
  Interventions: Drug: SI-B001; Drug: SI-B003

INTERVENTIONS:
Drug: SI-B001 — Administration by intravenous infusion
Drug: SI-B003 — Administration by intravenous infusion

SUMMARY:
Phase Ib: To observe the safety and tolerability of the combination of SI-B001 and SI-B003, and to determine the recommended dose of phase II clinical study (RP2D) in the indication of locally advanced or metastatic non-small cell lung cancer. Phase II: To evaluate the efficacy of SI-B001+SI-B003 combination with or without chemotherapy in patients with locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Subjects must agree to complete ctDNA testing during the screening period;
6. Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) patients;
7. Agree to provide archived or fresh tumor tissue samples from primary or metastatic lesions;
8. Must have at least one measurable lesion as defined by RECIST v1.1;
9. Performance status score: ECOG ≤1;
10. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
11. No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50%;
12. Organ function levels must meet the requirements without transfusion, albumin, colony-stimulating factors, any cell growth factors, and/or platelet-raising drugs within 14 days before the first dose of the study drug;
13. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
14. Urine protein ≤1+ or ≤1000 mg/24h;
15. Female subjects of childbearing potential or male subjects with partners of childbearing potential must use highly effective contraception from 7 days before the first dose until 24 weeks after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Prior to signing the informed consent form, relevant genetic alterations were indicated;
2. For patients enrolled in Phase II, any of the following conditions apply: a) Patients suitable for and willing to undergo local therapy; b) Patients who have received systemic chemotherapy;
3. Symptomatic brain parenchymal or leptomeningeal metastases, deemed ineligible by the investigator;
4. Participation in any other clinical trial within 4 weeks prior to the administration of this trial's investigational product (based on the last dose date);
5. Use of chemotherapy, biologic therapy, immunotherapy, etc., within 4 weeks or 5 half-lives prior to the first dose, or palliative radiotherapy, small-molecule targeted therapy, or other antitumor treatments within 2 weeks before the first dose;
6. Major surgery (as defined by the investigator) within 4 weeks prior to the first dose;
7. Requirement for systemic corticosteroids or immunosuppressive therapy within 2 weeks before the study drug administration;
8. Pulmonary diseases graded as ≥3 according to NCI-CTCAE v5.0; history of interstitial lung disease (ILD), current ILD, or suspected ILD during screening;
9. Concurrent pulmonary disease resulting in clinically significant respiratory impairment;
10. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening (excluding catheter-related thrombosis);
11. Active infection requiring intravenous anti-infective therapy;
12. Imaging findings indicating tumor invasion or encasement of major thoracic, cervical, or pharyngeal blood vessels, with a risk of bleeding post antitumor therapy;
13. Prior immunotherapy leading to ≥Grade 3 immune-related adverse events (irAE) or ≥Grade 2 immune-related myocarditis;
14. Use of live attenuated vaccines within 4 weeks before the first dose of the study drug;
15. Use of immunomodulatory drugs within 14 days before the first dose of the study drug;
16. Patients at risk of active autoimmune diseases or with a history of autoimmune diseases;
17. History of other malignancies within 5 years before the first dose;
18. Positive for human immunodeficiency virus (HIV) antibodies, active tuberculosis, active hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection;
19. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg);
20. History of severe cardiovascular or cerebrovascular diseases;
21. Patients with significant serous cavity effusion, symptomatic effusion, or poorly controlled effusion;
22. History of allogeneic stem cell, bone marrow, or organ transplantation;
23. History of hypersensitivity to recombinant humanized antibodies or any excipients of SI-B001 or SI-B003;
24. History of autologous or allogeneic stem cell transplantation;
25. Pregnant or lactating women;
26. Any other condition deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib/II: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of SI-B001+SI-B003.
Phase Ib/II: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Dose Limited Toxicity (DLT) | Up to approximately 24 months
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Phase Ib: Maximum Tolerated dose (MTD) or maximum administered dose (MAD) | Up to approximately 24 months
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.

SECONDARY OUTCOMES:
Phase Ib/II: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of SI-B001+SI-B003. The type, frequency and severity of TEAE will be evaluated during the treatment of SI-B001+SI-B003.
Phase Ib/II: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib/II: Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase Ib/II: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of SI-B001+SI-B003 to the first date of either disease progression or death, whichever occurs first.
Phase Ib/II: Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of SI-B001+SI-B003 will be investigated.
Phase Ib/II: Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of SI-B001+SI-B003 will be investigated.
Phase Ib/II: Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of SI-B001+SI-B003 prior to the next dose will be administered.
Phase Ib: T1/2 | Up to approximately 24 months
  Half-life (T1/2) of SI-B001+SI-B003 will be investigated.
Phase Ib: AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
Phase Ib: CL | Up to approximately 24 months
  The serum clearance rate of SI-B001+SI-B003 per unit time will be investigated.
Phase Ib/II: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-SI-B001, SI-B003 antibody (ADA) will be evaluated.
Phase Ib/II: Neutralizing antibody (Nab) | Up to approximately 24 months
  Incidence and titer of Nab of SI-B001 and SI-B003 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China